CLINICAL TRIAL: NCT05080075
Title: Platelet Rich Plasma in Knee Osteoarthritis: Establishing Clinical Guidelines to Predict and Maximize Outcomes
Brief Title: Platelet Rich Plasma in Knee Osteoarthritis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Christian Wuescher, Assistant Professor, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301106-UT
Record Dates: First submitted 2021-09-17; First posted 2021-10-15 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
Keywords: Platelet rich plasma; PRP; Knee osteoarthritis; Platelet concentration
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This study involves a single group, all of whom will be receiving the same treatment (platelet rich plasma injection into the knee)
Masking Description: All patients will get the treatment, and all those providing care and all involved in the study, including the research participants are aware of this
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants receiving a platelet rich plasma injection (Experimental): All patients in the study will be receiving a platelet rich plasma injection, and we will be following their clinical outcomes
  Interventions: Biological: Platelet Rich Plasma Injection

INTERVENTIONS:
Biological: Platelet Rich Plasma Injection — Research participants own blood will be used to prepare the platelet rich plasma injectate, which will be injected into the affected knee using ultrasound guidance.
  Other Names: PRP Injection

SUMMARY:
In this study, the investigators will be performing intra-articular platelet rich plasma (PRP) injections for patients experiencing pain related to osteoarthritis of the knee. The investigators will be following clinical outcomes, and how they relate to concentrations of the PRP samples as well as following opioid and emergency room utilization pre and post-injection.

DETAILED DESCRIPTION:
Osteoarthritis is the most common form of arthritis and results in pain and stiffness in the affected area and, depending on the joint, can lead to difficulty with mobility as well as with performing basic activities of daily living. Conservative management of this condition includes physical therapy, activity modification, bracing, medications, and corticosteroid injections. When conservative treatment measures have failed, patients are often left with a choice between surgery, specifically total knee arthroplasty, and long-term pain medications, including opioid medications. In the midst of the opioid epidemic, physicians are seeking non-opioid alternatives for treating pain when other conservative treatments have failed. One such alternative treatment option is an intraarticular platelet rich plasma (PRP) injection.

The goal of PRP is to stimulate the body's existing regenerative capabilities. Since it is known that platelets play a key role in the body's natural healing processes, multiple clinical trials have been conducted to determine if injecting the affected joint with a platelet rich sample of their own blood promotes healing and thus improves pain and function for patients suffering from osteoarthritis. The studies involving PRP have yielded some promising outcomes, however much remains unknown about maximizing outcomes using this technology and a clear and defined protocol for this intervention does not yet exist.

This study aims to clarify some of the factors that affect clinical outcomes, such as platelet and cell concentrations (both in a serum sample and in the centrifuged PRP sample) and patient demographics. Determining if higher platelet counts in the serum sample are associated with better outcomes could potentially be used to prognosticate patient outcomes and candidacy for the procedure. The investigators are examining if PRP injections reduce the costly utilization of emergency room care and use of opioid pain medications before and after the procedure. The investigators are correlating how specific PRP cell and substance concentrations (platelet, monocytes, etc.) affect clinical outcomes as well. Ultimately, our hope is that this study will contribute to the growing evidence that PRP is a safe and effective treatment option for debilitating knee osteoarthritis, that it can improve pain and function and reduce opioid use and emergency room utilization.

This study takes place at the University of Toledo Physical Medicine and Rehabilitation outpatient clinic. 50 subjects is the minimum required to answer the aims of this study but 100 will be the target number for this study over the course of one year. Members of the study will be recruiting patients by informing physicians in the area about the study and requesting referrals to the clinic for anyone that might meet criteria and expresses interest in the study (focusing on orthopaedics, rheumatology, internal medicine and family medicine). Study members will also be sending out brochures to inform local health care providers as well as the surrounding public about the study, and information on how to arrange a clinic visit to evaluate candidacy. Brochures may be sent in the form of paper copies, FAX or email with an attached brochure. Additionally, the investigators will be informing patients already established with providers from our clinics about the study. These patients may be contacted at any of the physicians' sites of service.

Patients meeting criteria, including documented knee osteoarthritis and associated pain, will have pre and post intra-articular PRP injection visits where information will be gathered for future analysis. The patient will initially be asked to come in to the Physical Medicine and Rehabilitation clinic after expressing interest in being a part of the study. During that initial visit, the patient will be given the initial screening form with inclusion criteria and exclusion criteria and it will be determined if they are a candidate for the study. If they do meet the criteria for inclusion, they will then be informed of the risks and benefits of the study as well as what would be required of them should they choose to enroll. The patient will then be given the consent form. If the patient signs the consent form and would like to join the study, the investigators will schedule a follow-up visit which will include the injection. At that visit, the patients who are physically able to bear children will be screened for pregnancy with a urine pregnancy test. Once the pregnancy tests are confirmed negative, they, along with all other patients, will be given the initial surveys to fill out including a review of their past medical history, the Visual Analog Scale (VAS) pain score questionnaire, and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire. Once the patients have filled these all out, they will undergo a blood draw of approximately 60 mL of their blood. Some of this sample will then be sent up to a lab where a complete blood count will be run. The remaining portion of the sample will be used for preparation of the platelet-rich plasma (PRP) using the Tortland Protocol developed by Paul Tortland, DO. After centrifugation, the PRP will be loaded into a syringe to be injected into the patient's knee. During preparation of the PRP, small samples will be obtained from the whole blood, PRP, and concentrated PRP while in the biosafety cabinet and analyzed for quantification of the cell types present and for characterization of the platelets (activation status, functionality assays). All immunology lab space stated on this protocol is BSL2 certified for use of untested human blood products. Once the concentrated PRP is obtained it will be brought back to the clinic for the injection.

While the patient is waiting for the platelet-rich plasma to be prepared, the Timed-Up-and-Go (TUG) test will be performed in the clinic to assess the patient's baseline functional ability prior to receiving the injection. Within 1 hour of the patient providing the sample of blood, the platelet-rich plasma sample will be brought back down from the lab. At that time, the patient will be brought to an exam room and the platelet-rich plasma injection will be performed on the affected knee under ultrasound-guidance. A trained physician will perform the injection using a 2.5 inch, 22-gauge needle and freeze spray will be used as a topical anesthetic for the 4-6 mL injection of platelet-rich plasma into the affected knee.

Post-procedure, the patient will be contacted to set-up a 4 week, 3 month, 6 month, and 1 year follow-up appointment at which time they will be brought back into the Physical Medicine and Rehabilitation clinic. At the 4 week appointment, the patient will be filling out a post-injection survey to explain if they experienced any adverse effects from the injection. In addition, the patient will have the opportunity at this appointment to ask any questions or voice any concerns that may have come up after the injection. At the 3 month, 6 month, and 1 year appointments, the patients will fill out post-injection surveys (Post-Injection Medical Survey) regarding Emergency Department and opioid medication utilization since the injection as well as updated VAS pain score and WOMAC questionnaires. The patient will also have the TUG test performed again during these appointments. After the 1 year follow-up, the patient will no longer be followed for purposes of this study. It is important to note that only treating physicians and nurses, medical students obtaining consent, and medical assistants rooming patients will see identifiable information. All other study related data or information will be de-identified using a number system. All study personnel will be informed that information, included protected health information, is confidential.

The results from the follow-up appointment will be compared to the patient's baseline results using the key code to match the de-identified information. These will results will all be compiled into the data collection spreadsheet. Descriptive statistics will be used to summarize the patients' clinical scores by demographic variables. Repeated measures ANOVA will be used to test for changes in VAS pain score, Timed Up and Go, Opioid utilization, Emergency Room Utilization and WOMAC questionnaires over time.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain or swelling that has been present for greater than 3 months
* Knee pain greater than or equal to 3 out of 10 on the visual analog scale
* Previous radiological evidence (X-ray) of osteoarthritis
* Age 18 or older

Exclusion Criteria:

* Unable to provide consent for enrollment in the study
* Unable to avoid NSAIDs during the study (must stop 7 days before injection)
* Age less than 18
* Confirmed rheumatologic disease affecting the knee
* Significant trauma to the knee within 2 months that resulted in pain and/or swelling
* Active malignancy
* Pregnancy
* Local injections to the knee within the last 3 months
* Previous knee surgery
* Other causes of knee pain (nerve pain, referred pain, infection of the knee joint, etc)
* History of platelet disorder
* History of thrombocytopenia
* History of severe anemia
* Severe cardiovascular disease
* Active infection
* Immunosuppression/immunodepression
* Currently taking anticoagulant/antiaggregant
* History of severe psychiatric disorder with psychosis
* Assistive device required for household ambulation within the previous 3 months
* Current IV drug user

Additionally this study requires that, for safety purposes, enrolled patients live within 2 hours driving distance from the study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Initial Pain outcomes | Start of the study, pre-injection
  The investigators will have patients rate pain levels using the visual analog scale (VAS), which measures pain on a 1-10 point scale. A score of 10 indicates the highest level of pain. These will be performed on the day of the platelet rich plasma injection, shortly before the procedure is performed.
Pain outcomes, 3 months | 3 months
  The investigators will have patients rate pain levels using the visual analog scale (VAS), which measures pain on a 1-10 point scale. A score of 10 indicates the highest level of pain.
Pain outcomes, 6 months | 6 months
  The investigators will have patients rate pain levels using the visual analog scale (VAS), which measures pain on a 1-10 point scale. A score of 10 indicates the highest level of pain.
Pain outcomes, 1 year | 1 year
  The investigators will have patients rate pain levels using the visual analog scale (VAS), which measures pain on a 1-10 point scale. A score of 10 indicates the highest level of pain.
Functional status outcomes using the Western Ontario and McMaster University Arthritis Index (WOMAC), initial | Start of the study, pre-injection
  Research participants will fill out a the WOMAC questionnaire. The WOMAC is a self administered questionnaire consisting of 24 items divided into subscales including pain (0-20), stiffness (0-8) and physical function (0-68). Higher scores indicate worse pain, stiffness and functional limitations.
Functional status outcomes using the Western Ontario and McMaster University Arthritis Index (WOMAC), 3 months | 3 months
  Research participants will fill out a the WOMAC questionnaire. The WOMAC is a self administered questionnaire consisting of 24 items divided into subscales including pain (0-20), stiffness (0-8) and physical function (0-68). Higher scores indicate worse pain, stiffness and functional limitations.
Functional status outcomes using the Western Ontario and McMaster University Arthritis Index (WOMAC), 6 months | 6 months
  Research participants will fill out a the WOMAC questionnaire. The WOMAC is a self administered questionnaire consisting of 24 items divided into subscales including pain (0-20), stiffness (0-8) and physical function (0-68). Higher scores indicate worse pain, stiffness and functional limitations.
Functional status outcome using the Timed up and go (TUG) test, initial | Start of the study, pre-injection
  The investigators will have participants perform a TUG test. The TUG test is an investigator administered test measuring the time it takes research participants to stand from a chair, walk three meters, turn around, walk back and sit down. It is timed in seconds, and a longer time to perform this task indicates a lower level of function.
Functional status outcome using the Timed up and go (TUG) test, 3 months | 3 months
  The investigators will have participants perform a TUG test. The TUG test is an investigator administered test measuring the time it takes research participants to stand from a chair, walk three meters, turn around, walk back and sit down. It is timed in seconds, and a longer time to perform this task indicates a lower level of function.
Functional status outcome using the Timed up and go (TUG) test, 6 months | 6 months
  The investigators will have participants perform a TUG test. The TUG test is an investigator administered test measuring the time it takes research participants to stand from a chair, walk three meters, turn around, walk back and sit down. It is timed in seconds, and a longer time to perform this task indicates a lower level of function.
Functional status outcome using the Timed up and go (TUG) test, 1 year | 1 year
  The investigators will have participants perform a TUG test. The TUG test is an investigator administered test measuring the time it takes research participants to stand from a chair, walk three meters, turn around, walk back and sit down. It is timed in seconds, and a longer time to perform this task indicates a lower level of function.
Correlation of outcomes with whole blood and platelet rich plasma (PRP) concentrations | Through study completion, 1 year
  The investigators will be determining if there is a correlation between the pain (VAS) and all functional outcomes (WOMAC and TUG) listed above, and whole blood and platelet rich plasma (PRP) concentrations. For PRP concentrations the investigators will be assessing platelet (and platelet activation), monocyte, neutrophil levels using flow cytometry. For whole blood concentrations the investigators will be using the hospitals lab system. These concentrations will be measured once on the day of the injection for each participant.

SECONDARY OUTCOMES:
Opioid utilization, initial | Start of the Study, pre-injection
  Research participants will fill out a questionnaire before the platelet rich plasma injection asking about opioid use prior to the injection. The questionnaire is titled "Pre-Injection Medical Survey" and asks a question regarding what medications are used to treat knee pain (opioids are included in this list)
Opioid utilization, 3 months | 3 months
  Research participants will fill out a questionnaire after the platelet rich plasma injection asking about opioid use after the injection. The questionnaire is titled "Post-Injection Medical Survey" and asks a question indicating whether or not the participant reduced their opioid use for knee pain following the injection.
Opioid utilization, 6 months | 6 months
  Research participants will fill out a questionnaire after the platelet rich plasma injection asking about opioid use after the injection. The questionnaire is titled "Post-Injection Medical Survey" and asks a question indicating whether or not the participant reduced their opioid use for knee pain following the injection.
Opioid utilization, 1 year | 1 year
  Research participants will fill out a questionnaire after the platelet rich plasma injection asking about opioid use after the injection. The questionnaire is titled "Post-Injection Medical Survey" and asks a question indicating whether or not the participant reduced their opioid use for knee pain following the injection.
Emergency room utilization, initial | Start of the study, pre-injection
  Research participants will fill out a questionnaire regarding emergency room utilization. The questionnaires are titled "Pre-Injection Medical Survey" and asks a questions regarding the number of emergency room visits the research participants have had for their knee pain
Emergency room utilization, 3 months | 3 months
  Research participants will fill out a questionnaire regarding emergency room utilization. The questionnaires is titled "Post-Injection Medical Survey" and asks a question regarding the number of emergency room visits the research participants have had since the injection
Emergency room utilization, 6 months | 6 months
  Research participants will fill out a questionnaire regarding emergency room utilization. The questionnaires is titled "Post-Injection Medical Survey" and asks a question regarding the number of emergency room visits the research participants have had since the injection
Emergency room utilization, 1 year | 1 year
  Research participants will fill out a questionnaire regarding emergency room utilization. The questionnaires is titled "Post-Injection Medical Survey" and asks a question regarding the number of emergency room visits the research participants have had since the injection
Correlation of outcomes and patient demographics and co-morbidities | Through study completion, 1 year
  The investigators will be determining if there is a correlation between clinical outcomes (pain scores (VAS) and functional measures (WOMAC and TUG) as described above) and patient demographics (Age, height/weight (BMI), gender, smoking history, alcohol history, allergies, race/ethnicity) as well as co-morbidities (diabetes, CKD, hypertension, COPD, CHF, CAD, peripheral vascular disease, anemia with hemoglobin < 9 in the previous 12 months). This information will be gathered by utilizing a self administered questionnaire prior to the injection, and then correlating outcomes to these demographics and co-morbidities. The questionnaire is titled "Pre-Injection Medical Survey"

CONTACTS AND LOCATIONS:
Overall Officials: Christian Wuescher, MD, Principal Investigator — University of Toledo; Ashley Schneider, MD, Study Director — University of Toledo; Leah Wuescher, PhD, Study Director — University of Toledo
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belk JW, Kraeutler MJ, Houck DA, Goodrich JA, Dragoo JL, McCarty EC. Platelet-Rich Plasma Versus Hyaluronic Acid for Knee Osteoarthritis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Am J Sports Med. 2021 Jan;49(1):249-260. doi: 10.1177/0363546520909397. Epub 2020 Apr 17. PMID 32302218
- [Background] Cole BJ, Karas V, Hussey K, Pilz K, Fortier LA. Hyaluronic Acid Versus Platelet-Rich Plasma: A Prospective, Double-Blind Randomized Controlled Trial Comparing Clinical Outcomes and Effects on Intra-articular Biology for the Treatment of Knee Osteoarthritis. Am J Sports Med. 2017 Feb;45(2):339-346. doi: 10.1177/0363546516665809. Epub 2016 Oct 21. PMID 28146403
- [Background] Dernek B, Kesiktas FN, Duymus TM, Aydin T, Isiksacan N, Diracoglu D, Aksoy C. Effect of platelet concentration on clinical improvement in treatment of early stage-knee osteoarthritis with platelet-rich plasma concentrations. J Phys Ther Sci. 2017 May;29(5):896-901. doi: 10.1589/jpts.29.896. Epub 2017 May 16. PMID 28603367
- [Background] Di Martino A, Di Matteo B, Papio T, Tentoni F, Selleri F, Cenacchi A, Kon E, Filardo G. Platelet-Rich Plasma Versus Hyaluronic Acid Injections for the Treatment of Knee Osteoarthritis: Results at 5 Years of a Double-Blind, Randomized Controlled Trial. Am J Sports Med. 2019 Feb;47(2):347-354. doi: 10.1177/0363546518814532. Epub 2018 Dec 13. PMID 30545242
- [Background] Filardo G, Di Matteo B, Di Martino A, Merli ML, Cenacchi A, Fornasari P, Marcacci M, Kon E. Platelet-Rich Plasma Intra-articular Knee Injections Show No Superiority Versus Viscosupplementation: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1575-82. doi: 10.1177/0363546515582027. Epub 2015 May 7. PMID 25952818
- [Background] Filardo G, Kon E, Pereira Ruiz MT, Vaccaro F, Guitaldi R, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma intra-articular injections for cartilage degeneration and osteoarthritis: single- versus double-spinning approach. Knee Surg Sports Traumatol Arthrosc. 2012 Oct;20(10):2082-91. doi: 10.1007/s00167-011-1837-x. Epub 2011 Dec 28. PMID 22203046
- [Background] Ghai B, Gupta V, Jain A, Goel N, Chouhan D, Batra YK. [Effectiveness of platelet rich plasma in pain management of osteoarthritis knee: double blind, randomized comparative study]. Braz J Anesthesiol. 2019 Sep-Oct;69(5):439-447. doi: 10.1016/j.bjan.2019.06.003. Epub 2019 Oct 28. PMID 31672420
- [Background] Gormeli G, Gormeli CA, Ataoglu B, Colak C, Aslanturk O, Ertem K. Multiple PRP injections are more effective than single injections and hyaluronic acid in knees with early osteoarthritis: a randomized, double-blind, placebo-controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Mar;25(3):958-965. doi: 10.1007/s00167-015-3705-6. Epub 2015 Aug 2. PMID 26233594
- [Background] Kon E, Buda R, Filardo G, Di Martino A, Timoncini A, Cenacchi A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma: intra-articular knee injections produced favorable results on degenerative cartilage lesions. Knee Surg Sports Traumatol Arthrosc. 2010 Apr;18(4):472-9. doi: 10.1007/s00167-009-0940-8. Epub 2009 Oct 17. PMID 19838676
- [Background] Lana JF, Macedo A, Ingrao ILG, Huber SC, Santos GS, Santana MHA. Leukocyte-rich PRP for knee osteoarthritis: Current concepts. J Clin Orthop Trauma. 2019 Oct;10(Suppl 1):S179-S182. doi: 10.1016/j.jcot.2019.01.011. Epub 2019 Jan 14. PMID 31700210
- [Background] Lin KY, Yang CC, Hsu CJ, Yeh ML, Renn JH. Intra-articular Injection of Platelet-Rich Plasma Is Superior to Hyaluronic Acid or Saline Solution in the Treatment of Mild to Moderate Knee Osteoarthritis: A Randomized, Double-Blind, Triple-Parallel, Placebo-Controlled Clinical Trial. Arthroscopy. 2019 Jan;35(1):106-117. doi: 10.1016/j.arthro.2018.06.035. PMID 30611335
- [Background] O'Connell B, Wragg NM, Wilson SL. The use of PRP injections in the management of knee osteoarthritis. Cell Tissue Res. 2019 May;376(2):143-152. doi: 10.1007/s00441-019-02996-x. Epub 2019 Feb 13. PMID 30758709
- [Background] Park YB, Kim JH, Ha CW, Lee DH. Clinical Efficacy of Platelet-Rich Plasma Injection and Its Association With Growth Factors in the Treatment of Mild to Moderate Knee Osteoarthritis: A Randomized Double-Blind Controlled Clinical Trial As Compared With Hyaluronic Acid. Am J Sports Med. 2021 Feb;49(2):487-496. doi: 10.1177/0363546520986867. PMID 33523756
- [Background] Patel S, Dhillon MS, Aggarwal S, Marwaha N, Jain A. Treatment with platelet-rich plasma is more effective than placebo for knee osteoarthritis: a prospective, double-blind, randomized trial. Am J Sports Med. 2013 Feb;41(2):356-64. doi: 10.1177/0363546512471299. Epub 2013 Jan 8. PMID 23299850
- [Background] Raeissadat SA, Rayegani SM, Babaee M, Ghorbani E. The effect of platelet-rich plasma on pain, function, and quality of life of patients with knee osteoarthritis. Pain Res Treat. 2013;2013:165967. doi: 10.1155/2013/165967. Epub 2013 Dec 9. PMID 24386565
- [Background] Rahimzadeh P, Imani F, Faiz SHR, Entezary SR, Zamanabadi MN, Alebouyeh MR. The effects of injecting intra-articular platelet-rich plasma or prolotherapy on pain score and function in knee osteoarthritis. Clin Interv Aging. 2018 Jan 4;13:73-79. doi: 10.2147/CIA.S147757. eCollection 2018. PMID 29379278
- [Background] Riboh JC, Saltzman BM, Yanke AB, Fortier L, Cole BJ. Effect of Leukocyte Concentration on the Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis. Am J Sports Med. 2016 Mar;44(3):792-800. doi: 10.1177/0363546515580787. Epub 2015 Apr 29. PMID 25925602
- [Background] Sanchez M, Fiz N, Azofra J, Usabiaga J, Aduriz Recalde E, Garcia Gutierrez A, Albillos J, Garate R, Aguirre JJ, Padilla S, Orive G, Anitua E. A randomized clinical trial evaluating plasma rich in growth factors (PRGF-Endoret) versus hyaluronic acid in the short-term treatment of symptomatic knee osteoarthritis. Arthroscopy. 2012 Aug;28(8):1070-8. doi: 10.1016/j.arthro.2012.05.011. PMID 22840987
- [Background] Simental-Mendia M, Vilchez-Cavazos JF, Pena-Martinez VM, Said-Fernandez S, Lara-Arias J, Martinez-Rodriguez HG. Leukocyte-poor platelet-rich plasma is more effective than the conventional therapy with acetaminophen for the treatment of early knee osteoarthritis. Arch Orthop Trauma Surg. 2016 Dec;136(12):1723-1732. doi: 10.1007/s00402-016-2545-2. Epub 2016 Aug 9. PMID 27506585
- [Background] Taniguchi Y, Yoshioka T, Kanamori A, Aoto K, Sugaya H, Yamazaki M. Intra-articular platelet-rich plasma (PRP) injections for treating knee pain associated with osteoarthritis of the knee in the Japanese population: a phase I and IIa clinical trial. Nagoya J Med Sci. 2018 Feb;80(1):39-51. doi: 10.18999/nagjms.80.1.39. PMID 29581613